CLINICAL TRIAL: NCT04913597
Title: A Prospective Observational Study of Switching Avatrombopag and Rh-TPO in Chinese Adult Patients With Primary Immune Thrombocytopenia
Brief Title: A Study of Switching Avatrombopag and Rh-TPO in ITP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Fuhaixia, associate chief physician, Peking University People's Hospital
Other Study IDs: ITP-SWITCH1
Record Dates: First submitted 2021-05-29; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Corticosteroid-resistant or Relapsed ITP
Keywords: Immune Thrombocytopenia; Recombinant human thrombopoietin; avatrombopag; switching
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recombinant human thrombopoietin (rh-TPO) group: Patients who fail previous steroids and avatrombopag and then switch to Rh-TPO will be enrolled. The reason for switch will be recorded. Patients will be given rh-TPO 300 U/kg once daily for 14 days as initial treatment. After initial treatment, maintenance therapy were performance. At initial therapy, rhTPO will be suspended when platelet counts ≥100×10^9 / L. During maintenance therapy, patients with platelet counts >150×10^9 / L will suspend treatment until platelet counts drop to ≤150×10^9 / L. Dosing interval will be prolonged when platelet count is ≥100×10^9 / L to ≤150×10^9 / L. Dose modification is not required when platelet count is ≥30×10^9 / L to <100×10^9 / L. The efficacy, safety, and patient/physician preference will be assessed.
- Avatrombopag group: Patients who fail previous steroids and rh-TPO and then switch to avatrombopag will be enrolled. The reason for switch will be recorded. Patients will be given avatrombopag 20mg once daily as initiate treatment, and adjust the dosage according to the count of platelets. The maximum dose of avatrombopag is 40mg daily.Avatrombopag will be terminated any time the platelet counts increased above 250×10^9/L. Dose adjustment of avatrombopag will be allowed to maintain platelet counts between 30×10^9/L and 150×10^9/L. The efficacy, safety, and patient/physician preference will be assessed.

SUMMARY:
Thrombopoietin receptor agonists (TPO-RAs) represent a highly effective and well-tolerated second-line ITP treatment that provides excellent responses.If there is cross-resistance between 2 drugs for the treatment of adult ITP is still unkonwn.The purpose of this study is to investigate the efficacy and safety of switching avatrombopag and rh-TPO in adults with ITP.

DETAILED DESCRIPTION:
Thrombopoietin Receptor Agonists (TPO-RAs) are novel treatments for patients with chronic Primary Immune Thrombocytopenia (ITP). According to the findings of mechanism-based studies, rhTPO competes with endogenous TPO for binding to TPO-R while avatrombopag has an additive effect with endogenous TPO, indicating that the treatment mechanism and side-effect profiles could be somewhat different between these drugs. If there is cross-resistance between 2 drugs for the treatment of adult ITP is still no answer. The purpose of this study is to investigate the efficacy and safety of switching avatrombopag and rh-TPO in adults with ITP.This is a non-interventional study. Patients who fail previous steroids and receive rh-TPO and then switch to avatrombopag or vice versa will be enrolled. The reason for switch will be recorded. The efficacy, safety, and patient/physician preference will be assessed and compared between the two agents.

ELIGIBILITY:
Inclusion Criteria:

1.18 years or older 2.Primary ITP 3.Failed initial glucocorticosteroid treatment, 4.Applying rhTPO or Eltrombopag as subsequent treatment 5.Switch from rh-TPO to eltrombopag or vice versa 6.Normal neutrophils 7.Available follow-up at least 6 weeks after switching

Exclusion Criteria:

1. HIV positive status, or active infection of HBV or HCV
2. Suffering from a serious or progressive disease, which, in the investigator's judgment, put the subject at undue risk for participation in this study (i.e. cancer or pre-cancer, immunocompromised, uncontrolled diabetes, epilepsy, severe cardio-cerebrovascular disease(s) (i.e. stroke, idiopathic aortic stenosis, aneurysm, hypertrophic obstructive cardiomyopathy, ischaemic heart disease, tachyarrhythmias, severe heart failure [classified as NYHA III-IV], severe lung dysfunctions, etc))
3. History of thrombosis plus two or more risk factors as defined in Caprini thrombosis risk assessment model
4. Lactating or pregnant women, or WOCBP who are unwilling to use highly effective contraceptive measures during the study period
5. Abnormal liver and renal functions: AST or ALT or total bilirubin ≥1.5 × ULN, and/or creatinine ≥176.8 μmol/L
6. Women of childbearing potential (WOCBP) that are pregnant or wish to become pregnant during the prospective phase of the study.
7. Other conditions which the investigator considers inappropriate for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ITP patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Initial response after switching | 4 weeks
  Rate of response at 4 weeks after switching from rhTPO to avatrombopag or vise versa

SECONDARY OUTCOMES:
Response rate at 12 weeks after switching | 12 weeks
  Rate of response at 12 weeks after switching from rhTPO to avatrombopag or vise versa
Initial response after switching according to the reasons of switching | 4 weeks
  Rate of response at 1 month after switching according to the reasons of switching,such as lack of efficacy, Platelet count fluctuations, development of adverse events,patient's or doctor's preference
Rate of response at 12 weeks after switching according to the reasons of switching | 12 weeks
  Rate of response at 12 weeks after switching according to the reasons of switching,such as lack of efficacy, Platelet count fluctuations, development of adverse events,patient's or doctor's preference
Time to response | 4 weeks
  Time to CR or R from switching
Durable response | 24 weeks
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 24 weeks follow-up.
Incidence of bleeding events | 24 weeks
  Incidence of clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale
Immune Thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) | 24 weeks
  In all participants ,use ITP-PAQ to assess the Health Related Quality of Life(HRQoL) before and after treatment.
Functional Assessment of Chronic Illness Therapy fatigue subscale (FACIT-F) | 24 weeks
  In all participants ,use FACIT-F to assess the Health Related Quality of Life(HRQoL) before and after treatment.
Safety assessment | 24 weeks
  Number of Participants with side effects of the drugs

CONTACTS AND LOCATIONS:
Overall Officials: Haixia Fu, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neunert C, Terrell DR, Arnold DM, Buchanan G, Cines DB, Cooper N, Cuker A, Despotovic JM, George JN, Grace RF, Kuhne T, Kuter DJ, Lim W, McCrae KR, Pruitt B, Shimanek H, Vesely SK. American Society of Hematology 2019 guidelines for immune thrombocytopenia. Blood Adv. 2019 Dec 10;3(23):3829-3866. doi: 10.1182/bloodadvances.2019000966. PMID 31794604
- [Background] Liu XG, Bai XC, Chen FP, Cheng YF, Dai KS, Fang MY, Feng JM, Gong YP, Guo T, Guo XH, Han Y, Hong LJ, Hu Y, Hua BL, Huang RB, Li Y, Peng J, Shu MM, Sun J, Sun PY, Sun YQ, Wang CS, Wang SJ, Wang XM, Wu CM, Wu WM, Yan ZY, Yang FE, Yang LH, Yang RC, Yang TH, Ye X, Zhang GS, Zhang L, Zheng CC, Zhou H, Zhou M, Zhou RF, Zhou ZP, Zhu HL, Zhu TN, Hou M. Chinese guidelines for treatment of adult primary immune thrombocytopenia. Int J Hematol. 2018 Jun;107(6):615-623. doi: 10.1007/s12185-018-2445-z. Epub 2018 Apr 4. PMID 29619624
- [Background] Provan D, Arnold DM, Bussel JB, Chong BH, Cooper N, Gernsheimer T, Ghanima W, Godeau B, Gonzalez-Lopez TJ, Grainger J, Hou M, Kruse C, McDonald V, Michel M, Newland AC, Pavord S, Rodeghiero F, Scully M, Tomiyama Y, Wong RS, Zaja F, Kuter DJ. Updated international consensus report on the investigation and management of primary immune thrombocytopenia. Blood Adv. 2019 Nov 26;3(22):3780-3817. doi: 10.1182/bloodadvances.2019000812. PMID 31770441
- [Background] Wormann B. Clinical indications for thrombopoietin and thrombopoietin-receptor agonists. Transfus Med Hemother. 2013 Oct;40(5):319-25. doi: 10.1159/000355006. Epub 2013 Sep 11. PMID 24273485
- [Background] Bussel JB. Avatrombopag. Br J Haematol. 2018 Nov;183(3):342-343. doi: 10.1111/bjh.15568. Epub 2018 Oct 23. No abstract available. PMID 30351482
- [Background] Kuter DJ. The biology of thrombopoietin and thrombopoietin receptor agonists. Int J Hematol. 2013 Jul;98(1):10-23. doi: 10.1007/s12185-013-1382-0. Epub 2013 Jul 3. PMID 23821332